CLINICAL TRIAL: NCT05981807
Title: Prevalence of Genital, Anal and Oral HPV Infection and Sexually Transmitted Infections, and of Anal Dysplasia in the Transgender Population (PrevHPV-TG)
Brief Title: HPV Infection, Sexually Transmitted Infections and Anal Dysplasia in the Transgender Population
Acronym: PrevHPV-TG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-A00672-43
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Human Papillomavirus Infection; Human Immunodeficiency Virus Infection; Sexually Transmitted Diseases
Keywords: HPV; HIV; Transgender; Dysplasia; Neisseria gonorrhoeae; Chlamydia trachomatis; Syphilis; STI
MeSH Terms: conditions — Papillomavirus Infections; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Syphilis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transgender population: Cohort of transgender people (man to woman and woman to man)

SUMMARY:
The goal of this observational study is to estimate the prevalence of HPV infections anal and ENT level and according to HIV status in transgender (TG) population. The main question it aims to answer is:

* What is the prevalence of HPV lesions in transgender population (TG);
* What kind of high risk HPV (hrHPV) and low risk HPV (lrHPV) are detected at the genital, anal and ENT level

DETAILED DESCRIPTION:
Context:

The few publications with an individualized transgender (TG) population have been conducted in South America (Peru, Argentina) showing very high anal or ano-genital hrHPV prevalences of around 97% (dos Ramos Farias et al., 2011; Brown et al., 2016). Recently a study conducted in 22 TGs showed a high prevalence of anal dysplastic lesions with low grade lesions detected in 8 individuals and high grade in 3 individuals (Kobayashi et al., 2017). Thus, in the face of this high prevalence of 50% anal dysplasia, the TG population therefore appears to be at risk for developing anal dysplastic lesions and this needs to be explored in another TG population. Furthermore, to our knowledge, no study has evaluated the concomitant prevalence of hrHPV infection at the anogenital and ENT levels in the transgender population. The Infectious and Tropical Diseases Department of Bichat-Claude Bernard Hospital is particularly involved in the follow-up of transgender individuals with a large active file that participates in clinical research projects (Pommier et al., 2019; Bertin et al., 2019; Phung et al., 2018).

Objectives:

Principal objective The primary objective of this study is to determine the prevalence of HPV lesions in transgender population (TG).

Secondary objectives

Secondary objectives include:

1. Estimate the prevalence of HPV infections at the genital, anal and ENT level and according to HIV status;
2. To estimate the prevalence of hrHPV infections at the genital, anal and ENT levels, globally and according to HIV status;
3. To estimate the prevalence of lrHPV infections at the genital, anal and ENT level globally and by HIV status;
4. Describe the types of hrHPV and lrHPV detected at the genital, anal and ENT level;
5. To estimate the prevalence of dysplastic lesions (low grade and high grade) by HIV status;
6. To estimate the prevalence of bacterial Sexually Transmitted Infections (STIs): Neisseria gonorrhoeae, Chlamydia trachomatis and Syphilis, globally and by anatomical site and HIV status.

Methodology This is a national, non-interventional, cross-sectional, monocentric study among TG people (man to woman, and woman to man)

Estimated enrolment 200 participants

Outcomes Primary outcome:

The prevalence of HPV infections among TG people. Prevalence is defined as the percentage of subjects with HPV infection among TG people included, regardless the site where infection was detected.

Secondary outcomes:

1. The prevalence of HPV infections in each anatomical site (genital, anal and ENT) and by HIV status.
2. The prevalence of hrHPV infections in each anatomical site (genital, anal and ENT), globally and according to HIV status.
3. The prevalence of lrHPV infections in each anatomical site (genital, anal and ENT), globally and by HIV status.
4. The types of hrHPV and lrHPV in each anatomical site (genital, anal).
5. The prevalence of dysplastic lesions (low grade and high grade) by HIV status.
6. The prevalence of bacterial STIs: Neisseria gonorrhoeae, Chlamydia trachomatis and Syphilis, globally, by anatomical site and HIV status.

Eligibility Inclusion criteria

* Age ≥ 18 years
* To belong to transgender population : i.e. people who doesn't identify to the gender assigned at birth
* To be affiliated to a social security system or be beneficiary of the Aide Médicale d'Etat (AME)

Non-inclusion criteria

* To have ever been vaccinated against HPV
* Research participation refusal
* People under guardianship or curatorship, or deprived of liberty by administrative or judiciary measure

Statistical methods Individuals' characteristics will be described for all included subjects. Continuous variables will be described using mean, standard deviation, median, interquartiles values, minimal and maximal values. Qualitative variables will be described using numbers and percentages by modality. Prevalences will be described by proportion and their confidence interval will be calculated under binomial law. All statistical tests will be performed using 5% as significance level. Prevalence of high risk HPV infection in each anatomical site and the concordance of HPV types by anatomical site will be determined using Fleiss Kappa test.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* To belong to transgender population : i.e. people who doesn't identify to the gender assigned at birth
* To be affiliated to a social security system or be beneficiary of AME

Exclusion criteria:

* To have ever been vaccinated against HPV
* Research participation refusal
* People under guardianship or curatorship, or deprived of liberty by administrative or judiciary measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include people who belong to the transgender population : i.e. people who do not identify to the gender assigned at birth (man to woman and woman to man).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HPV infection in transgender population | 12 months
  The prevalence of HPV infections is defined as the percentage of subjects with HPV infection among transgender people included, regardless the site of infection.

SECONDARY OUTCOMES:
Prevalence of HPV infections at the genital, anal and ENT level and according to HIV status | 12 months
  We will estimate the prevalence of HPV infections in each anatomical site (genital, anal and ENT) and according to HIV status.
Prevalence of hrHPV infections at the genital, anal and ENT levels, globally and according to HIV status | 12 months
  We will estimate the prevalence of hrHPV infections in each anatomical site (genital, anal and ENT), globally and according to HIV status.
Prevalence of lrHPV infections at the genital, anal and ENT level globally and by HIV status | 12 months
  We will estimate the prevalence of lrHPV infections in each anatomical site (genital, anal and ENT), globally and by HIV status.
Types of hrHPV and lrHPV detected at the genital, anal and ENT level | 12 months
  We will describe the types of hrHPV and lrHPV detected at the genital, anal and ENT level
Prevalence of dysplastic lesions (low grade and high grade) by HIV status | 12 months
  We will estimate the prevalence of dysplastic lesions (low grade and high grade) by HIV status.
Prevalence of bacterial sexually transmitted infections: Neisseria gonorrhoeae, Chlamydia trachomatis and Syphilis, globally and by anatomical site and HIV status | 12 months
  We will estimate the prevalence of bacterial sexually transmitted infections: Neisseria gonorrhoeae, Chlamydia trachomatis and Syphilis, globally, by anatomical site and HIV status.

CONTACTS AND LOCATIONS:
Overall Officials: Jade GHOSN, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris